CLINICAL TRIAL: NCT05666817
Title: The Effect of Postpartum Breastfeeding Education Given to Women Who Had Normal Vaginal and Cesarean Delivery on Breastfeeding Self-efficacy and Breastfeeding Success
Brief Title: The Effect of Postpartum Breastfeeding Education on Breastfeeding Self-efficacy and Breastfeeding Success
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Nur Bahar Kuru Aktürk, STUDENT, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: p8v6z463
Record Dates: First submitted 2022-12-19; First posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Breastfeeding
Keywords: Breastfeeding; Breastfeeding Education; Self-Efficacy; Successful Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: The study will be conducted with 76 women, 38 controls and 38 interventions.
Who Masked: Participant
Masking Description: 2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experiment group (Experimental): Breastfeeding training will be given to each mother in the room she stays in the form of lectures and after the training, the question and answer method will be used. In addition, the practices explained by the researcher (the way of holding the baby, grasping the breast and positioning the baby appropriately for the baby, determining the position suitable for breastfeeding and the process of expressing and storing breast milk) will be demonstrated using the mother demonstration method in order to evaluate whether the mother understands the breastfeeding education after the breastfeeding training. Breastfeeding training will take approximately 40-45 minutes.
  Interventions: Other: breastfeeding education
- Control group (No Intervention): No attempt will be made to the mothers in the control group following the pre-test application, within the scope of the post-test application before discharge; Breastfeeding Knowledge Level Diagnostic Form, LATCH Scale and Postnatal Self-Efficacy Scale will be applied. In addition to the breastfeeding education given to the intervention group following the post-test application to the mothers in the control group, a guide on the importance of breast milk and breastfeeding will also be given.

INTERVENTIONS:
Other: breastfeeding education — Mothers in the intervention group will be given breastfeeding training after the pre-test application. The content of breastfeeding education is as follows;
  * General information about breastfeeding,
  * General information about breast milk and the benefits of breast milk,
  * Benefits of breastfeeding for mother and baby,
  * How the baby should be held during breastfeeding, the baby's position,
  * Effective breastfeeding positions for the mother,
  * Ensuring that the baby holds the breast correctly,
  * Providing the correct breastfeeding technique,
  * Breast milking and storage conditions,
  * The necessity and benefits of continuing breastfeeding.
  Arms: experiment group

SUMMARY:
Objective: This study will be conducted as a pre-test post-test randomized controlled study in order to determine the effect of postpartum breastfeeding education given to women who had normal vaginal delivery and cesarean section on breastfeeding self-efficacy and breastfeeding success.

Materials and Methods: The data of the study were collected with "Descriptive Information Form, Breastfeeding Knowledge Level Diagnosis Form, LATCH Breastfeeding Diagnosis and Evaluation Scale and Postpartum Breastfeeding Self-Efficacy Scale". SPSS 25.0 (Statistical Package for Social Science) program will be used in the analysis of the data.

Design: Randomized controlled.

The study included 76 women who had normal vaginal and cesarean delivery and met the inclusion criteria (Research Research group, 38 control group) in Zeynep Kamil Gynecology and Pediatrics Education and Hospital Postpartum Postpartum Postpartum Service in Istanbul.

DETAILED DESCRIPTION:
Breast milk is a newborn-specific food that varies according to the baby's needs, body weight and the density that the baby can digest. Breastfeeding, on the other hand, is the most natural action that allows mother's milk to meet with the newborn. In addition to providing benefits for the growth and development of the baby, it contributes significantly to the maintenance of general health in advanced ages, the improvement of health and the reduction of the effect of risk factors affecting health. The concept of breastfeeding self-efficacy is the mother's perception of breastfeeding. Self-efficacy perception about breastfeeding determines the behavior of mothers to continue breastfeeding, whether they can cope with breastfeeding problems, their thoughts and attitudes about breastfeeding. Mother's age, education level, baby's weight and mother's number of births are concepts that can affect breastfeeding self-efficacy perception. Although there are many studies on breastfeeding in the literature, a limited number of studies have been found that determine the effect of the early results of postpartum breastfeeding education on breastfeeding self-efficacy and breastfeeding success.

This study aims to determine the effect of postpartum breastfeeding education given to women who had normal vaginal and cesarean delivery on breastfeeding self-efficacy and breastfeeding success.

The objectives of the research;

* To determine the effect of postpartum breastfeeding education given to women with normal vaginal delivery on breastfeeding self-efficacy.
* To determine the effect of postpartum breastfeeding education given to women who had cesarean section on breastfeeding self-efficacy.
* To determine the effect of postpartum breastfeeding education given to women who had normal vaginal delivery on breastfeeding success.
* To determine the effect of postpartum breastfeeding education given to women who had cesarean section on breastfeeding success.

ELIGIBILITY:
Inclusion Criteria:

* The following criteria will be taken into account for the individuals to be included in the intervention and control groups:

  * Volunteering to participate in the research (Annex-1),
  * Being between the ages of 18-40,
  * Ability to read and write,
  * Being able to read and understand Turkish,
  * Not having a hearing, speaking or visual impairment,
  * Having had a normal or cesarean delivery,
  * Having a live birth and having a healthy baby.

Exclusion Criteria:

* Women under 18 years of age, • Women whose babies were taken to the neonatal intensive care unit.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2022-12-10 (Actual); Primary Completion 2022-12-18 (Actual); Study Completion 2022-12-18 (Actual)

PRIMARY OUTCOMES:
Introductory Information Form | 5 minute
  This form; mother's age, education status, social security, economic status, number of pregnancies, gestational week, type of delivery, baby's gender, desire for pregnancy, how many times she applied to a health institution during her pregnancy, which health institution she applied to for control, the status of receiving breastfeeding training during pregnancy, If she received breastfeeding training, from whom she received it, the status of reading magazines/brochures about breastfeeding during pregnancy, and the status of wanting to receive free breastfeeding training after delivery.

SECONDARY OUTCOMES:
Breastfeeding Knowledge Level Diagnosis Form | 10 minute
  This form, which was prepared by the researcher in order to measure breastfeeding efficiency; It consists of 15 questions about breastfeeding initiation time, breast milk storage conditions, breastfeeding positions, breastfeeding duration and frequency, general information about breastfeeding and breast milk. Each question has three options: yes, no and I don't know. 1 point is given for each correct answer, and 0 points are given for incorrect and I don't know. The questions in the form are mixed right and wrong. If questions 1, 2, 3, 4, 5, 6, 9, 10, 11, 12, 14, 15 are marked as correct, and questions 7, 8, and 13 as incorrect, the highest total score that can be obtained from the form will be 15.

OTHER OUTCOMES:
LATCH Scale | 10 minute
  This scale is a diagnostic method created in 1986 to evaluate breastfeeding success, whose scoring system is similar to the APGAR scoring system. The application time takes about 5-8 minutes. This diagnostic and evaluation scale has been developed to provide an objective diagnosis and evaluation of breastfeeding, to evaluate the breastfeeding success of the mother, to create a common language for health professionals and to be used in scientific studies.
Postnatal Self-Efficacy Scale | 10 minute
  Developed by Dennis in 2003, this scale consists of 14 items. The scale assesses how competent mothers feel about breastfeeding. The fourteen-item scale includes a 5-point Likert-type assessment consisting of "Not at all sure: 1, Not quite sure: 2, Sometimes sure: 3, Sure: 4, Very sure: 5".

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Akturk NBK, Kolcu M. The effect of postnatal breastfeeding education given to women on breastfeeding self-efficacy and breastfeeding success. Rev Assoc Med Bras (1992). 2023 Aug 21;69(8):e20230217. doi: 10.1590/1806-9282.20230217. eCollection 2023. PMID 37610927